CLINICAL TRIAL: NCT03514433
Title: Translating Research Into Practice: A Regional Collaborative to Reduce Disparities in Breast Cancer Care
Brief Title: Translating Research Into Practice: Patient Navigation for Breast Cancer
Acronym: TRIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Boston University (Other); University of Massachusetts, Worcester (Other); Beth Israel Deaconess Medical Center (Other); Tufts Medical Center (Other); Dana-Farber Cancer Institute (Other); Massachusetts General Hospital (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-37314; 1U01TR002070-01 (NIH)
Record Dates: First submitted 2018-04-21; First posted 2018-05-02 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Cancer, Breast
Keywords: Patient Navigation; Disparity; Social Determinants
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: A randomized cluster stepped wedge design will be conducted. This pragmatic design involves a sequential, randomized roll-out of the intervention across 5 participating clinical sites or "clusters" over 3 month intervals or "steps". Consistent with a stepped wedge design with one cluster per step, prior to the collection of data in the pre-intervention period, the investigators will generate a set of uniform random numbers for each of the five clusters to assign a starting period for the study intervention. There will be no crossover of patients from usual care to the intervention. That is, patients at each site during the pre-intervention period will experience only usual care and will act as historical controls and those enrolled after the initiation of intervention will experience the intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control- Usual Care (No Intervention): This study will be utilizing electronic health record data to identify patients that match the TRIP eligibility criteria and received patient navigation prior to study rollout. These patients will receive standard patient navigation at their care site and will act as controls in comparison to the TRIP experimental group.
- TRIP Patient Navigation Intervention (Experimental): This study will be enhancing current patient navigation at the participating 5 hospitals with the 3 components of the TRIP intervention (a shared patient registry, a social determinants of health platform, and additional training and support for Patient Navigators). All patients that are identified as TRIP eligible will receive these intervention benefits and will be categorized into the experimental arm of the study.
  Interventions: Other: TRIP Patient Navigation Intervention

INTERVENTIONS:
Other: TRIP Patient Navigation Intervention — The TRIP intervention will replace the current standard of care at the 5 participating hospitals once it is rolled out on-site. Any TRIP eligible patients receiving patient navigation services over the course of the study will receive the enhanced services.
  Arms: TRIP Patient Navigation Intervention

SUMMARY:
The TRIP Project aims to overcome barriers to widespread implementation and dissemination of evidence-based practices that will improve the delivery of guideline-concordant care to vulnerable women with breast cancer. To accomplish this goal the study team will create (a) regional patient registries; (b) systematic screening for social barriers to care with a personalized referral plan; and (c) patient navigation services that integrate into one model of care to improve the quality and effectiveness of care delivery, for minority and/or low-income women with breast cancer in Boston.

DETAILED DESCRIPTION:
This community-engaged program will demonstrate the feasibility of community-academic partnerships to provide innovations in information sharing and systems implementation targeted to reduce treatment disparities. Patient navigators will be able to utilize the patient database to track their patients throughout their treatment, and receive guidance regarding recommended social resources to patients experiencing hardships via the social determinants platform.

Who: The four Massachusetts Clinical and Translational Science Award (CTSA) hubs (Boston University, Harvard University, Tufts University, and University of Massachusetts) partnered with the Boston Breast Cancer Equity Coalition, and the 5 hospitals that care for women with breast cancer.

Patient population: about 1,300 vulnerable inner city women with risk for delay in breast cancer care. Massachusetts (MA) Cancer Registry data identified the following characteristics of Boston residents with greatest delays in breast cancer treatment: Black, Hispanic, non-English speaking, and public health insurance. Five health care institutions care for >90% of these women:

1. Beth Israel Deaconess Medical Center (site PI: Ted James, MD)
2. Boston Medical Center (PI: Tracy Battaglia MD, MPH)
3. Brigham Women's Hospital/Dana-Farber Cancer Institute (PI: Jennifer Haas MD, MPH)
4. Massachusetts General Hospital (site PI: Beverly Moy, MD)
5. Tufts Medical Center (PI: Karen Freund MD, MPH)

University of Massachusetts Medical Center (PI: Stephenie Lemon, PhD) will play an integral role in the planning and implementation of the TRIP intervention but is not a clinical site.

ELIGIBILITY:
Inclusion Criteria:

1. are an adult female 18 years of age or older;
2. reside within 25 miles of the City of Boston;
3. have any of the following risk factors for delays in care: are Black and/or Hispanic ethnicity, do not speak English as their primary language, and/or have only public insurance or are uninsured at the time of diagnosis.

Exclusion Criteria:

1. cancer diagnosis made > 60 days prior to enrollment, such that the ability of the intervention to effect the outcome is limited;
2. presence of a cognitive impairment such as dementia or delirium from any cause (e.g. metabolic, medication or drug induced), given the unique challenges to their treatment decision making/ adherence and the fact that the intervention would not include the patient directly, but rather the family;
3. home residence is outside of the city of Boston, Massachusetts.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All women with breast cancer diagnosed at a participating study site during the study period will be eligible for inclusion if they meet three study criteria
Enrollment: 1725 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Battaglia, MD., MPH, Principal Investigator — Boston Medical Center
Locations (5):
- United States (5):
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available. Participant data will be shared after de-identification and only through aggregate form through publications. Supporting documentation such as the study protocol will be available for review. Data dictionaries are available upon reasonable request.

REFERENCES:
- [Derived] Rajabiun S, Xiao V, Bak S, Robbins C, Casanova N, Cabral HJ, Lemon SC, Haas JS, Freund KM, Battaglia T; TRIP Consortium. Using community-engaged methods to develop a study protocol for a cost analysis of a multi-site patient navigation intervention for breast cancer care. BMC Health Serv Res. 2022 Jul 8;22(1):881. doi: 10.1186/s12913-022-08192-y. PMID 35804359
- [Derived] Loo S, Mullikin K, Robbins C, Xiao V, Battaglia TA, Lemon SC, Gunn C; TRIP Consortium. Patient navigator team perceptions on the implementation of a citywide breast cancer patient navigation protocol: a qualitative study. BMC Health Serv Res. 2022 May 21;22(1):683. doi: 10.1186/s12913-022-08090-3. PMID 35597947
- [Derived] LeClair AM, Battaglia TA, Casanova NL, Haas JS, Freund KM, Moy B, Parsons SK, Ko NY, Ross J, Ohrenberger E, Mullikin KR, Lemon SC. Assessment of patient navigation programs for breast cancer patients across the city of Boston. Support Care Cancer. 2022 Mar;30(3):2435-2443. doi: 10.1007/s00520-021-06675-y. Epub 2021 Nov 12. PMID 34767089

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants are newly diagnosed breast oncology patients at one of the five participating clinical sites. Over 18 months in a stepped wedge design sites were randomized to the time they began to implement the intervention, with a new site initiating the intervention about every 3 months. Control- Usual Care data from each serves as the comparison.
Groups:
- Sequence 1 (Hospital 1): Sequence: 22 months of Usual Care, 2 months of implementation, then 38 months of Intervention Control (Usual Care): These patients will receive standard patient navigation at their care site and will act as controls in comparison to the TRIP experimental group.
  Intervention: This study will be enhancing current patient navigation at the participating 5 hospitals with the 3 components of the TRIP intervention (a shared patient registry, a social determinants of health platform, and additional training and support for Patient Navigators). All patients that are identified as TRIP eligible will receive these intervention benefits and will be categorized into the experimental arm of the study.
  TRIP Patient Navigation Intervention: The TRIP intervention wilt replace the current standard of care at the 5 participating hospitals once it is rolled out on-site. Any TRIP eligible patients receiving patient navigation services over the course of the study will receive the enhanced services.
- Sequence 2 (Hospital 2): Sequence: 25 months of Usual Care, 2 months of implementation, then 35 months of intervention.
  Control (Usual Care): These patients will receive standard patient navigation at their care site and will act as controls in comparison to the TRIP experimental group.
  Intervention: This study will be enhancing current patient navigation at the participating 5 hospitals with the 3 components of the TRIP intervention (a shared patient registry, a social determinants of health platform, and additional training and support for Patient Navigators). All patients that are identified as TRIP eligible will receive these intervention benefits and will be categorized into the experimental arm of the study.
  TRIP Patient Navigation Intervention: The TRIP intervention wilt replace the current standard of care at the 5 participating hospitals once it is rolled out on-site. Any TRIP eligible patients receiving patient navigation services over the course of the study will receive the enhanced services.
- Sequence 3 (Hospital 3): Sequence: 28 months of Usual Care, 2 months of implementation, then 32 months of intervention.
  Control (Usual Care): These patients will receive standard patient navigation at their care site and will act as controls in comparison to the TRIP experimental group.
  Intervention: This study will be enhancing current patient navigation at the participating 5 hospitals with the 3 components of the TRIP intervention (a shared patient registry, a social determinants of health platform, and additional training and support for Patient Navigators). All patients that are identified as TRIP eligible will receive these intervention benefits and will be categorized into the experimental arm of the study.
  TRIP Patient Navigation Intervention: The TRIP intervention wilt replace the current standard of care at the 5 participating hospitals once it is rolled out on-site. Any TRIP eligible patients receiving patient navigation services over the course of the study will receive the enhanced services.
- Sequence 4 (Hospital 4): Sequence: 31 months of Usual Care, 2 months of implementation, then 29 months of intervention.
  Control (Usual Care): These patients will receive standard patient navigation at their care site and will act as controls in comparison to the TRIP experimental group.
  Intervention: This study will be enhancing current patient navigation at the participating 5 hospitals with the 3 components of the TRIP intervention (a shared patient registry, a social determinants of health platform, and additional training and support for Patient Navigators). All patients that are identified as TRIP eligible will receive these intervention benefits and will be categorized into the experimental arm of the study.
  TRIP Patient Navigation Intervention: The TRIP intervention wilt replace the current standard of care at the 5 participating hospitals once it is rolled out on-site. Any TRIP eligible patients receiving patient navigation services over the course of the study will receive the enhanced services.
- Sequence 5 (Hospital 5): Sequence: 36 months of Usual Care, 2 months of implementation, then 24 months of intervention.
  Control (Usual Care): These patients will receive standard patient navigation at their care site and will act as controls in comparison to the TRIP experimental group.
  Intervention: This study will be enhancing current patient navigation at the participating 5 hospitals with the 3 components of the TRIP intervention (a shared patient registry, a social determinants of health platform, and additional training and support for Patient Navigators). All patients that are identified as TRIP eligible will receive these intervention benefits and will be categorized into the experimental arm of the study.
  TRIP Patient Navigation Intervention: The TRIP intervention wilt replace the current standard of care at the 5 participating hospitals once it is rolled out on-site. Any TRIP eligible patients receiving patient navigation services over the course of the study will receive the enhanced services.
Period: Usual Care
Arm/Group | Sequence 1 (Hospital 1) | Sequence 2 (Hospital 2) | Sequence 3 (Hospital 3) | Sequence 4 (Hospital 4) | Sequence 5 (Hospital 5)
Started | 111 | 38 | 177 | 83 | 141
Completed | 111 | 38 | 177 | 83 | 141
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Intervention
Arm/Group | Sequence 1 (Hospital 1) | Sequence 2 (Hospital 2) | Sequence 3 (Hospital 3) | Sequence 4 (Hospital 4) | Sequence 5 (Hospital 5)
Started | 317 | 75 | 372 | 144 | 267
Completed | 317 | 75 | 372 | 144 | 267
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- TRIP Patient Navigation Intervention: This study will be enhancing current patient navigation at the participating 5 hospitals with the 3 components of the TRIP intervention (a shared patient registry, a social determinants of health platform, and additional training and support for Patient Navigators). All patients that are identified as TRIP eligible will receive these intervention benefits and will be categorized into the experimental arm of the study.
  TRIP Patient Navigation Intervention: The TRIP intervention will replace the current standard of care at the 6 participating hospitals once it is rolled out on-site. Any TRIP eligible patients receiving patient navigation services over the course of the study will receive the enhanced services.
- Total: Total of all reporting groups
Arm/Group | Control- Usual Care | TRIP Patient Navigation Intervention | Total
Number analyzed (Participants) | 550 | 1175 | 1725
Age, Customized [Count of Participants; unit: Participants]
  <50 years | 132 | 293 | 425
  50-64 years | 213 | 483 | 696
  65+ years | 205 | 399 | 604
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 550 | 1175 | 1725
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 127 | 296 | 423
  Nonhispanic White | 91 | 236 | 327
  Nonhispanic Black | 243 | 483 | 726
  Nonhispanic Asian | 70 | 129 | 199
  Other | 4 | 18 | 22
  Missing or Unknown | 15 | 13 | 28
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 550 | 1175 | 1725

OUTCOME MEASURES:

1. Primary Outcome: Time-to-treatment Post-diagnosis
Description: The receipt of care will be defined as initiation of care within 365 days. This will be a continuous outcome defined as the number of days from definitive tissue biopsy (Time 0) to treatment initiation (Time 1). Treatment initiation is defined as the date of first cancer treatment: surgical, radiation, or systemic therapy (including chemotherapy, immunotherapy, targeted therapy, hormonal therapy). Time to treatment initiation can take any value from 0 days to 365 days (study period). The clinical outcome will be derived from data in the patient's medical record.
Time Frame: Within 365 days of enrollment
Population: Data were available for 529 of the 550 controls and 1151 of the 1175 participants in the intervention group.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control- Usual Care | TRIP Patient Navigation Intervention
Number analyzed (Participants) | 529 | 1151
days | 44.78 (39.54) | 45.40 (33.98)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Control- Usual Care | TRIP Patient Navigation Intervention
All-Cause Mortality (participants affected / at risk) | 14/550 | 16/1175
Serious Adverse Events (participants affected / at risk) | 0/550 | 0/1175
Other Adverse Events (participants affected / at risk) | 0/550 | 0/1175

LIMITATIONS AND CAVEATS:
Generalizability was limited since participants were only enrolled within the Boston health systems with existing navigation. In addition, the COVID-19 pandemic caused care disruption.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT03514433/Prot_SAP_001.pdf
  • Informed Consent Form (2019-11-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT03514433/ICF_000.pdf